CLINICAL TRIAL: NCT05498727
Title: Assessing the Effectiveness of Integration of Rapid Antigen Testing for SARS-CoV-2 in MNCH, HIV and TB Services in Cameroon and Kenya: A Pre- and Post- Implementation Evaluation (Effectiveness Study)
Brief Title: Evaluation of the Integration of Ag-RDTs for COVID-19 in MNCH, HIV and TB Services in Cameroon and Kenya
Status: Completed | Type: Observational
Sponsor: Elizabeth Glaser Pediatric AIDS Foundation (Other)
Collaborators: UNITAID (Other); Kenya Ministry of Health (Other Government); Ministry of Public Health, Cameroon (Unknown)
Responsible Party: Sponsor
Other Study IDs: EG0276
Record Dates: First submitted 2022-08-10; First posted 2022-08-12 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2024-01

CONDITIONS: COVID-19
Keywords: Antigen rapid diagnostic test; Integration; COVID-19; Health Facilities; Africa; Effectiveness
MeSH Terms: conditions — COVID-19 | interventions — Seroconversion

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Maternal Newborn and Child Health (MNCH) Clinics: Clients attending for routine service delivery at MNCH clinics.
  Interventions: Diagnostic Test: Integration of SARS-CoV 2 Testing in HIV, MNCH and TB Clinics
- HIV Clinics: Patients attending for HIV clinic services
  Interventions: Diagnostic Test: Integration of SARS-CoV 2 Testing in HIV, MNCH and TB Clinics
- Tuberculosis (TB) Clinics: Patients attending TB clinic services.
  Interventions: Diagnostic Test: Integration of SARS-CoV 2 Testing in HIV, MNCH and TB Clinics

INTERVENTIONS:
Diagnostic Test: Integration of SARS-CoV 2 Testing in HIV, MNCH and TB Clinics — This study employs a quasi-experimental pre-and-post SARS-CoV-2 Ag-RDT integration design in all facilities implementing the 61 facilities in Cameroon and Kenya in Cameroon and Kenya.

SUMMARY:
In many national Coronavirus Disease 2019 (COVID-19) response plans, including in Kenya and Cameroon, antigen detection tests are being used to improve access for Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) testing. Targeting the populations most at risk for COVID-19 disease, including pregnant women, people living with HIV, and patients with tuberculosis (TB), and those who are the most vulnerable to transmission to other populations, can reduce the negative impact of the SARS-CoV-2 pandemic. Catalyzing COVID-19 Action (CCA) aims to strengthen detection by screening and diagnosing cases of SARS-CoV-2 in MNCH clinics, HIV clinics, and TB clinics and enhancing the management of COVID-positive cases. The main goal of the CCA project is to reduce deaths and severe illnesses caused by COVID-19 through early access to reliable diagnosis and effective treatment through innovative models of care. Both countries will conduct a pre- and post-implementation evaluation to compare screening, testing, care, and treatment of patients undergoing COVID-19 screening, testing, and treatment before and after the integration of facilities taking part in the CCA project.

DETAILED DESCRIPTION:
Background The use of simple and affordable rapid diagnostic antigen detection tests (Ag-RDT) to expand access to Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) testing is being incorporated into many national Coronavirus Disease 2019 (COVID-19) response plans, including in Cameroon and Kenya. Ag-RDT are less expensive, highly sensitive, provide faster results, and require little technical support to diagnose SARS-CoV-2 infection. Targeting populations at high risk for COVID-19 and severe outcomes, and at risk of transmitting infection to other vulnerable populations has the potential to mitigate the propagation and effects of the SARS-CoV-2 pandemic. These high-risk populations include pregnant women, people living with HIV, and patients with tuberculosis. Data on SARS-CoV-2 infection in these populations in Africa and on the integration of Ag-RDT testing into Maternal Neonatal and Child Health (MNCH), HIV, and TB clinics are limited.

Objectives The main objective of this study is to evaluate the effectiveness of the integration of SARS-CoV-2 Ag-RDT in the MNCH, HIV and TB clinics in Cameroon and Kenya on SARS-CoV-2 testing and routine service delivery as compared to baseline. Investigators will also describe facility and individual factors that are associated with SARS-CoV-2 infection and the cascade of care and clinical outcomes in the post -integration period.

Methods A pre- and post-implementation evaluation design will be implemented in both countries to compare COVID-19 testing before and after the Ag-RDT integration. The study will be conducted in 61 purposively selected facilities (31 in Kenya and 30 in Cameroon). The population will include attendees at the MNCH, HIV and TB clinics at all the 61 facilities. SARS-CoV-2 screening will be performed for all attendees and testing offered to those who meet eligibility criteria as part of the MOH supported COVID-19 response. The study will consist of abstraction/extraction of routine facility service delivery records for secondary analysis of the program data only. There is no specific sample size but investigators estimate >10,000 clinic attendees will be screened.

Study Outcome The evidence generated by this evaluation will be used to support policy recommendations for improving COVID-19 testing, isolation, and treatment solutions in existing health platforms. This evaluation will allow for dissemination of results and subsequent adoption of proven models for integration and decentralization of COVID testing in multiple countries.

ELIGIBILITY:
Inclusion Criteria:

* MNCH services: all pregnant and breastfeeding women coming for antenatal care or post-natal care will be offered SARS-CoV-2 screening and testing; all children > 2 years brought to the facility for routine immunization or under 5 years old clinics and their mother or caregivers will also be offered this service.
* HIV services: all children (2-17 years) and adults (>18 years) attending HIV services, including those coming for a clinical or laboratory visit, those coming to collect medications or for counseling/support groups, and those who are accompanying patients (such as caregivers of HIV infected child, etc.) will be offered SARS-CoV-2 screening and testing.
* TB services: all children (2-17 years) and adults (>18 years) attending TB services, including those coming for a clinical or laboratory visit, those coming to collect medications or for TB preventive therapy, and those who are accompanying patients (such as parent of a child, household contact, etc).

Exclusion Criteria:

* Clinic attendees from MNCH, HIV and TB clinics who tested positive for SARS-CoV-2 within the past two weeks.

Min Age: 2 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: The population will include attendees at the MNCH, HIV and TB clinics at all of the CCA project sites in Cameroon and Kenya. SARS-CoV-2 screening and testing will be offered to all attendees per the eligibility criteria below.
Sampling Method: Non-Probability Sample
Enrollment: 527184 (Actual)
Dates: Start 2022-05-02 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Proportion of pediatric and adult clinic attendees tested for SARS-CoV-2 | Study evaluation period (9 months)
  Total number of clinic attendees tested with Ag-RDTs divided by the total number of clinic attendees
SARS-CoV-2 detection rate | Study evaluation period (9 months)
  Number of Ag-RDTs testing SARS-CoV-2 positive attendees divided by total number of clinic attendees multiplied by 100 (#SARS-CoV-2 infections detected per 100 clinic attendees).
Effect of integrated SARS-CoV-2 Ag-RDT testing on routine service delivery indicators | Study evaluation period (9 months)
  Comparison of corresponding monthly number of clinic attendees pre/post integration of Ag-RDTs into routine clinic services by taking a ratio of the total attendance and plotting the ratio over time

SECONDARY OUTCOMES:
Factors associated with proportion of clinic attendees screened and tested with SARS-CoV-2 Ag-RDT, linked to care and treatment among the attendees following the integration of SARS-CoV-2 Ag-RDT in MNCH, HIV and TB clinics. | Study evaluation period (9 months)
  Facility-level factors; facility level (hospital/health center/service entry points), location (region), support type, associated with screening and testing
Individual-level factors associated with SARS-CoV-2 infection, disease status, and outcomes | Study evaluation period (9 months)
  Distribution of client/patient demographic and clinical characteristics will be examined stratified by infection status using frequencies and proportion or means/medians as appropriate

CONTACTS AND LOCATIONS:
Overall Officials: Nilesh Bhatt, MD, PhD, Principal Investigator — Elizabeth Glaser Pediatric AIDS Foundation; Rose Otieno Masaba, MD, MSc, Principal Investigator — Elizabeth Glaser Pediatric AIDS Foundation; Boris Tchounga, MD, PhD, Principal Investigator — Elizabeth Glaser Pediatric AIDS Foundation
Locations (2):
- Health facilities in Cameroon, Yaoundé, Cameroon
- Health facilities in Kenya, Nairobi, Kenya

IPD SHARING:
Plan to Share IPD: Yes
Anonymized participant data will be made available upon requests directed to the corresponding author. Proposals will be reviewed and approved by the sponsor, investigator, and collaborators on the basis of scientific merit. After approval of a proposal, data can be shared through a secure online platform after signing a data-sharing agreement. All data will be made available for a minimum of 3 years from the end of the trial.
Supporting Information: Study Protocol
Time Frame: All data will be made available for a minimum of 3 years from the end of the trial.
Access Criteria: For any data request reach out the study protocol Principal Investigator (nbhatt@pedaids.org)

REFERENCES:
- [Derived] Tchounga BK, Hoffman N, Masaba R, Djikeussi T, Ndimbii J, Moma E, Pearson S, Sikuku E, Gitau V, Argaw S, Tchendjou P, Siamba S, Kimani N, Zoung-Kanyi Bissek AC, Fokam J, Tiam A, Yemaneberhan A, Guay L, Bhatt NB, Machekano R. Integrating SARS-CoV-2 rapid antigen testing in maternal, neonatal and child health, HIV, and TB clinics in Kenya and Cameroon: outcomes from the Catalysing COVID-19 Action Project. BMJ Public Health. 2024 Aug 8;2(Suppl 1):e001015. doi: 10.1136/bmjph-2024-001015. eCollection 2024 Jul. PMID 41221322